CLINICAL TRIAL: NCT00200824
Title: Effects of Soy Isoflavones on the Prostate, Breast and Bone
Brief Title: Effects of Soy Compounds on Breast Cancer, Prostate Cancer, and Bone Health
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: R01AT000486 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2006-08

CONDITIONS: Breast Cancer; Prostate Cancer
Keywords: isoflavones; soy; postmenopausal; men; prostate; breast; bone
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Multiple Endocrine Neoplasia Type 1

INTERVENTIONS:
Drug: Soy Isoflavone Nutritional Supplements

SUMMARY:
This study will determine the effects of soy products on in vitro surrogate cancer markers as well as bone density markers and quality of life parameters in men and women. This study will also determine concentrations of isoflavones (naturally occurring plant compounds that act like estrogen in the body) in prostate tissue that has been removed during prostatectomy, as well as in the blood.

DETAILED DESCRIPTION:
In the United States, consumption of soy products has dramatically increased in the past several years. Foods made from soy are high in isoflavones and evidence suggests that these isoflavones, genistein in particular, have many beneficial properties such as alleviating menopausal side effects and reducing the risk of osteoporosis, breast cancer, and prostate cancer. However, this data has been derived largely from studies with animal or cell models; human trials are limited. This study will determine the effects of soy isoflavones on quality of life and cancer and bone density markers.

While isoflavones have been purported to inhibit the proliferation of cancer cells, the concentrations required for this anti-cancer effect were determined to be much higher than the concentrations that can be achieved in plasma after intake of isoflavones. Recent animal studies have suggested that isoflavones may be concentrated 10-fold in tissue compared to blood concentrations. If this is true, then the higher concentration would be in the range found in the cancer cell line research to be protective of cancer. This study will determine whether tissue concentrations are similar to, higher than, or different than blood concentrations.

This study will last 5 years and will comprise three populations: men with prostate cancer on androgen ablation therapy, postmenopausal women on hormone replacement therapy (HRT), and postmenopausal women not on HRT. Participants will be randomly assigned to receive either isoflavone or placebo for two to four weeks. Participants' serum and serum extracts will be incubated with cultured human cell lines (prostate cancer, breast cancer and osteoblasts) and estrogenic and non-estrogenic mechanisms of action investigated. The human sera data will be complemented by parallel studies of direct addition of crystalline isoflavones (genistein, daidzein and equol) to the same cultured human cell lines. Participant's serum and urine also will be tested for markers of bone resorption and formation. Quality of life issues will be assessed with questionnaires.

ELIGIBILITY:
Inclusion Criteria

* Scheduled for prostatectomy
* Willing and able to consume study tablets for at least 2 weeks prior to surgery
* Willing to accept random assignment
* Signed informed consent

Exclusion Criteria

* Unwilling to avoid soy intake during the study period
* Currently taking antibiotics

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-05; Study Completion 2005-01

PRIMARY OUTCOMES:
Markers of Bone Density
Basic Science (e.g., proliferation of cancer cells in vitro)

SECONDARY OUTCOMES:
Bioavailability

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Gardner, Principal Investigator — Stanford University
Locations (1):
- Christopher Gardner, Stanford, California, United States